CLINICAL TRIAL: NCT01734564
Title: Phase II Study With Hiltonol and Dendritic Cells in Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-2010-01
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2016-05

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — poly ICLC; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hiltonol and autologous dendritic cells (Experimental): Hiltonol and autologous dendritic cells
  Interventions: Biological: Hiltonol and autologous dendritic cells
- Hiltonol, dendritic cells and radiation (Experimental): Hiltonol, dendritic cells and radiation.
  Interventions: Radiation: Hiltonol, dendritic cells and radiation

INTERVENTIONS:
Biological: Hiltonol and autologous dendritic cells — Hiltonol and autologous dendritic cells
  Arms: Hiltonol and autologous dendritic cells
Radiation: Hiltonol, dendritic cells and radiation — Hiltonol, autologous dendritic cells and radiation therapy. Radiation therapy will pursue an abscopal effect.
  Arms: Hiltonol, dendritic cells and radiation

SUMMARY:
In this phase II study, patients with solid tumors will receive treatment with hiltonol and autologous dendritic cells.

DETAILED DESCRIPTION:
In this phase II study, patients with solid tumors will receive treatment with intratumoral hiltonol and two cycles of autologous dendritic cells loaded with autologous tumor and administered subcutaneously. A new cohort will explore the role of radiation therapy, looking for an abscopal effect.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of advanced solid tumors
* Measurable disease
* Performance status 0, 1 or 2.
* Adequate renal, hepatic and bone marrow function
* Availability of tumor tissue, for maturing dendritic cells

Exclusion Criteria:

* Clinically relevant diseases or infections.
* concurrent participation in other clinical trial or administration or other antitumoral treatment
* Concurrent cancer, with the exceptions allowed by the PI.
* Pregnant or breast feeding women
* immunosuppressant treatment
* known uncontrolled central nervous system metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Response rate | 8-10 weeks

SECONDARY OUTCOMES:
Safety (Common Toxicity Criteria 4.0) | 8-10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jose Luis Perez Gracia, MD, PhD, Principal Investigator — Clinica Universidad de Navarra
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain